CLINICAL TRIAL: NCT07016009
Title: Randomized Controlled Trial of the Thrive Person-Centered Planning Program for Young Adults With FASD
Brief Title: Thrive Person-Centered Planning Program for Young Adults With Fetal Alcohol Spectrum Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Christie Petrenko, Associate Professor of Pediatrics, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00010579; 1R61AA030780 (NIH)
Record Dates: First submitted 2025-06-02; First posted 2025-06-11 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Fetal Alcohol Spectrum Disorders
Keywords: fetal alcohol spectrum disorders; person-centered planning
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thrive Program (Experimental)
  Interventions: Behavioral: Thrive Program
- Waitlist Comparison Group (No Intervention)

INTERVENTIONS:
Behavioral: Thrive Program — Thrive is a person-centered planning intervention that is based on self-determination theory and integrates elements of social network interventions. The proposed Thrive intervention has four phases: 1) Strengths & Network Assessment, 2) Network Engagement, 3) Goal Setting & Planning, and 4) Plan Implementation & Monitoring. It involves about 10-13 sessions and is delivered by a trained facilitator over Zoom.
  Arms: Thrive Program

SUMMARY:
This study is testing a new program called Thrive. The Thrive program was developed for young adults with fetal alcohol spectrum disorders (FASD). Thrive uses a person-centered planning approach, which means it focuses on what is most important to the young adult with FASD. The young adult invites people that support them to help them make plans to meet their goals. 60 young adults with FASD will participate in this study. Half of the young adults will try out the Thrive program immediately. The other half will be on a waitlist and will get to start the program about 8 months later. Everyone completes online surveys at three times during the study. They do surveys at the beginning of the study, after 4 months, and after 8 months. The goal of the study is to test if the Thrive program helps young adults meet their goals and get support when they need it.

DETAILED DESCRIPTION:
This type 1 hybrid effectiveness-implementation trial proposes a 2-arm parallel pilot RCT design. A total of 60 young adults with FASD will be randomly assigned into the (1) Thrive intervention or the (2) waitlist comparison group using a 50:50 allocation ratio. As this is a type 1 hybrid trial, measurement emphasizes effectiveness outcomes, with collection of some implementation outcomes/process to inform planning of subsequent larger scale community trials. Consistent with the pilot RCT design, analysis will focus on determining feasibility of the intervention, trial procedures and measurement, and intervention process. This information will optimize success of the planned R01 larger-scale RCT.

ELIGIBILITY:
Inclusion Criteria:

* Young adult between the ages of 18 and 25
* Lives in the United States
* Has a diagnosis of fetal alcohol spectrum disorder or confirmed prenatal alcohol exposure

Exclusion Criteria:

* Does not have access to the internet or data plan allowing video conferencing
* Is not able to listen or speak in English

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Group mean differences on Personal Well-being Index | Baseline to 8 months
  Participants will complete the Personal Well-being Index (PWI) at all time-points. The PWI is a brief measure of quality of life. The 8-item measure asks how people feel about their material, physical, mental, and general well-being. The Intellectual Disability Version uses more concrete item wording and a 5-point visual scale. Ratings are summed and higher scores reflect better perceived well-being. An effect size of 0.2 is small, 0.5 is medium, and 0.8 is large.
Group mean differences on Basic Psychological Need Satisfaction and Frustration Scale | Baseline to 8 months
  Participants will complete the Basic Psychological Need Satisfaction and Frustration Scale (BPNSF) at all timepoints. The BPNSF is a 24-item scale assessing both satisfaction and frustration relating to the three basic psychological needs identified in self-determination theory: autonomy, competence, and relatedness. Items are rated on a 5 point visual scale. Higher scores reflect greater need satisfaction.
Group mean differences on Medical Outcomes Study: Social Support Survey | Baseline to 8 months
  Participants will complete the Medical Outcomes Study: Social Support Survey (MOS-SSS) at all time-points. The MOS-SSS is a 19-item measure of perceived availability of social support including emotional, informational, tangible, positive social interaction, and affectionate sources of support. Higher scores reflect higher levels of perceived support.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes